CLINICAL TRIAL: NCT02712489
Title: A Roll-over Observational Study for the Extended Follow-up of the Volunteers of the ISS T-003 Trial (ISS T-003 EF-UP)
Brief Title: A Roll-over Observational Study for the Extended Follow-up of the Volunteers of the ISS T-003 Trial
Acronym: ISST-003EF-UP
Status: Completed | Type: Observational
Sponsor: Barbara Ensoli, MD, PhD (Other)
Collaborators: Italian Ministry of Foreign Affairs - General Direction for Cooperation and Development (Unknown)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Director National Aids Center, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS T-003 EF-UP
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: HIV Infections
Keywords: HAART-treated participants; Tat; Therapeutic immunization
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: All patients that participated to the therapeutic phase II trial of the Tat vaccine "ISS T-003"
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
A roll-over observational study (ISS T-003 EF-UP) is being conducted to extend the follow-up of the volunteers of the ISS T-003 trial in order to evaluate the persistence of vaccine immunogenicity as well as of the immunological and virological effects induced by the therapeutic immunization with Tat.

DETAILED DESCRIPTION:
An open label, non-interventional study roll-over study (ISS T-003 EF-UP) is being conducted to follow-up the persistence of vaccine humoral responses as well as of the immunological and virological effects induced by the therapeutic immunization with Tat.To this aim volunteers of the ISS T-003 study are included in one year study, with visits at weeks 0 and 24 and 54.

To assess the anti-Tat humoral immune response by the determination and titration of IgM, IgG and IgA anti-Tat antibodies (primary endpoint) and to evaluate CD4+ T cell counts and HIV-1 plasma viraemia (as secondary endpoint).

In addition, depending on the availability of residual specimens (PBMC, serum and plasma), further laboratory tests (i.e. HIV DNA copies in blood) to investigate in-depth the immunological and virological profile of the volunteers is being performed.

Physical examination is being performed to monitor the clinical status of the volunteers and to record the appearance of clinical signs and symptoms of disease progression as well as AIDS-defining events, data or records related to ARV treatment compliance. Pregnancy onset for female participants will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* previous participation in the ISS T-003 trial without withdrawal of consent;
* availability to participate in the extended follow-up study;
* signed informed consent.

Exclusion Criteria:

* The absence of any of the above criteria will exclude the participants from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HAART-treated patients who participated to the therapeutic phase II trial of the Tat vaccine "ISS T-003"
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Presence of specific anti-Tat humoral immune response | Through study completion, an average of 1 year
  anti-Tat IgM, IgG, IgA antibodies

SECONDARY OUTCOMES:
CD4+ T cell counts | Through study completion, an average of 1 year
HIV-1 RNA Viral Load | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Matsontso Mathebula Mecru Clinical Research Unit, Sefako Makgatho, Health Sciences University,, Medunsa, Gauteng, South Africa

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- See also: related info — http://www.hiv1tat-vaccines.info